CLINICAL TRIAL: NCT06999876
Title: The Effect of Combined Transcranial Pulse Current Stimulation (tPCS) and Transcutaneous Electrical Nerve Stimulation (TENS) on Lower Limb Motor Function in Subacute to Chronic Stroke Patients With Hemiplegia: A Double-blind, Sham-controlled, Randomized Controlled Study
Brief Title: The Effect of Combined Transcranial Pulse Current Stimulation (tPCS) and Transcutaneous Electrical Nerve Stimulation (TENS) on Lower Limb Motor Function in Subacute to Chronic Stroke Patients With Hemiplegia (COMPENSATOR-Stroke)
Acronym: COMPENSATOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, JING MINGXUE, Dr Jing Mingxue (Principal Investigator), National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-3371
Record Dates: First submitted 2025-05-13; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Stroke Patients With Hemiplegia or Hemiparesis in the Subacute Stage
Keywords: Transcranial Pulsed Current Simulation; Transcutaneous Electrical Nerve Stimulation; Lower limb motor function recovery; Spasticity; Gait dysfunction; Standing balance; Ambulation; Stroke; Hemiplegia; Hemiparesis
MeSH Terms: conditions — Muscle Spasticity; Stroke; Hemiplegia; Paresis

STUDY DESIGN:
Intervention Model Description: Active tPCS + TENS treatment (Intervention arm) This group will receive active TENS treatment delivered through Channel 2, 3 and 4 of The AscenZ-VIII Stimulator via 6*9cm Silica gel electrodes on top of the tPCS that is delivered through Channel 1. The placement of the electrodes will be on the part of the spinal segment innervating the lower limbs (L1-L5), the adductor muscles and the gastrocnemius muscles.
  Sham tPCS + TENS treatment (Control arm) Sham tPCS current will be delivered through Channel 1, while active TENS treatment delivered through Channel 2, 3 and 4 of The AscenZ-VIII Stimulator via surface electrodes. The placement of electrodes will be exactly the same as the active tPCS montage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Active tPCS + TENS treatment
  Interventions: Device: The AscenZ-VIII Stimulator (Investigational Medical Device)
- Control arm (Sham Comparator): Sham tPCS + TENS treatment
  Interventions: Device: The AscenZ-VIII Stimulator (Investigational Medical Device)

INTERVENTIONS:
Device: The AscenZ-VIII Stimulator (Investigational Medical Device) — Sham tPCS current will be delivered through Channel 1, while active TENS treatment delivered through Channel 2, 3 and 4 of The AscenZ-VIII Stimulator via surface electrodes. The placement of electrodes will be exactly the same as the active tPCS montage.
  Arms: Control arm
Device: The AscenZ-VIII Stimulator (Investigational Medical Device) — This group will receive active TENS treatment delivered through Channel 2, 3 and 4 of The AscenZ-VIII Stimulator via 6*9cm Silica gel electrodes on top of the tPCS that is delivered through Channel 1. The placement of the electrodes will be on the part of the spinal segment innervating the lower limbs (L1-L5), the adductor muscles and the gastrocnemius muscles.
  Arms: Intervention Arm

SUMMARY:
The goal of this study is to evaluate the effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in lower limb motor function recovery in stroke patients with hemiplegia or hemiparesis in the subacute stage.The main questions it aims to answer are:

Primary objective - To evaluate the effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in lower limb motor function recovery, in stroke patients with hemiplegia or hemiparesis in the subacute stage

Secondary Objectives -

1. To evaluate the effects of high frequency tPCS + TENS in treatment of lower limb spasticity related to stroke.
2. To evaluate the effects of high frequency tPCS + TENS in gait function improvement post stroke, including walking speed, mobility, balance and walking endurance.
3. To evaluate the effects of high frequency tPCS on pain, mood and QOL.

Researchers will compare the effects of high frequency tPCS + TENS to a control group which involves intervention with Sham device stimulation + TENS.

Participants will:

* Be identified, recruited and have baseline assessments during screening period
* First undergo a mandatory 2-hour device training at Visit 2 to ensure device competence.
* Proceed with up to 7 days of habituation for device use and tolerability.
* Carry out daily intervention sessions of 30 minutes for 30 days at home or inpatient setting.
* Phone call follow-up (Telephone/ Video Call Interview) 2 weeks post intervention
* Clinic visit at day 30 post intervention with allowance of + 7 days for study assessments
* Clinic visit at day 90 post intervention with allowance of +/- 7 days for study assessments
* Update study coordinators via messaging platforms with regards to device issues, adverse events, any other reporting or questions

DETAILED DESCRIPTION:
In this prospective, double-blind, sham-controlled randomized control study, a total of 90 participants with hemiplegia or hemiparesis post stroke will be recruited from National University Hospital (NUH) and Alexandra Hospital (AH) inpatient wards and outpatient clinic. 45 participants will be randomized to the intervention arm (Intervened with tPCS + TENS) and 45 participants will be randomized to the control arm (Sham device stimulation + TENS).

The study will consist of a Screening period of up to 14 days. Participants who fulfil all the inclusion criteria will be consented and recruited during this screening period, constituting as Visit 1 (Recruitment). During this visit, PI/ Co-I obtaining consent will ensure that patient/ caregiver meets the following criteria:

1. For patients where the caregiver is administering the treatment, study team will ensure that they are the primary caregiver of the patient.
2. Patient/ caregiver must be comfortable and committed in following directions for device usage.
3. Patient/ caregiver must not have mental disability.

After confirmation of the above criteria, patient/ caregiver will undergo a 2-hour hands-on training at NUH by trained study team.

A set of training slides titled "AscenZ-VIII User training slides" that is adapted from the standard "Instruction Manual AscenZVIII" will be utilized for the training session for patient/ caregiver. After which, a checklist titled "Home Training Checklist" will be completed by both the trainer and patient/caregiver. This checklist is aimed to ensure that all necessary components of training have been covered by the trainer and also for trainers to indicate confidence of patient/ caregiver during the training before both trainer and patient/ caregiver signs as a form of training acknowledgement.

Post training, a copy of the standard "Instruction Manual AscenZVIII" will be given to patient/ caregiver. Study team will emphasize to patient/ caregiver that they can contact study team at any juncture where they need additional clarifications relating to the device.

Depending on the hospitalization status at time of screening, the patient will be seen in the inpatient ward or specialist outpatient clinic at day 14 which is considered as Visit 2 (Randomization with allowance + 3 days). Allowance of up to 3 days is given in the event day 14 falls on a weekend/long weekend. Following Visit 2 (Randomization with allowance + 3 days), up to 3 days of habituation for device use and tolerability will take place. Participants will be required to receive the intervention at low levels of intensity to allow conditioning for the habituation period. Because of the nature of the intervention, it may cause some discomfort to the participants, hence conditioning will increase the tolerability of the treatment for the participants.

Intervention with tPCS will take place over 30 days either in the inpatient setting of NUH and AH or in the home setting, while the rehabilitation therapy sessions with physiotherapy and occupational therapy happening concurrently as per existing clinical treatment protocol. Treatment with tPCS and TENS will consist of a daily session of 30 minutes for 30 days. Compliance will be checked by research assistant via telephone or video call interview at regular interval. One group will be randomised to the sham device stimulation + TENS (Control) arm and one group will be randomised to the active device intervention arm (intervened with tPCS + TENS). The sham device stimulation (Control) arm have electrode placement in the exact manner as the treatment arm but receive very little transcranial stimulation such that the output is negligible.

Assessment will be done at the time of recruitment which constitutes as Visit 1 (Recruitment), and again at the Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days) and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).

Activities and assessments that are done under research activities include:

Visit 1 (Recruitment)

* Eligibility screening
* Consent taking
* Blood Pressure (Research procedure if not done clinically)
* Standard physio and occupational therapy sessions as prescribed by patient's physician (Research procedure if not done clinically)
* Stroke deficit scale (Baseline mRS, NIHSS)
* Clinical measures on lower limb motor function (Lower Extremity - Fugl Meyer Assessment Baseline, Time UP and Go Baseline, 6 Minute Walk Test Baseline, 10 Meter Walk Test Baseline)
* Clinical measures on lower limb spasticity - Hip, Knee Flexion, Ankle Flexor, Plantar (Modified Ashworth Scale Baseline, Modified Tardieu Scale Baseline)
* Balance (Berg Balance Scale Baseline)
* Pain (Pain Numeric Rating Scale Baseline)
* Mood (Hospital Anxiety and Depression Scale Baseline)
* FIM
* EQ5D-5L Baseline
* Overall length of stay in hospital
* Outcomes events/Complications

Visit 2 (Randomization with allowance of + 3 days):

* Randomization
* Commence first day of habituation, up to 3 days

Follow-up Telephone/ Video Call Interview, at 2 weeks post intervention (Research procedure)

- Patients will be asked regarding: i) Device related side-effects ii) Hospital re-admissions iii) Changes in medications iv) Device management (eg. Difficulties faced while using the device, Device working condition Damage to device, Device parts that require replacement, Re-supply of consumables, etc)

Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days):

* Treatment group OR Control Group - 30min daily for 30 days
* Stroke deficit scale (mRS, NIHSS)
* Clinical measures on lover limb motor function (Lower Extremity - Fugl Meyer Assessment, Time Up and Go, 6 Minute Walk Test, 10 Meter Walk Test )
* Clinical measures on lower limb spasticity - Hip, Knee Flexion, Ankle Flexor, Plantar (Modified Ashworth Scale, Modified Tardieu Scale)
* Balance (Berg Balance Scale)
* Pain (Pain Numeric Rating Scale)
* Mood (Hospital Anxiety and Depression Scale)
* FIM
* EQ5D-5L
* Overall length of stay in hospital
* Outcomes events/Complications

Visit 4 (Final follow-up, Day 90 post intervention with allowance of +/- 7 days):

* Stroke deficit scale (mRS, NIHSS)
* Clinical measures on lower limb motor function (Lower Extremity - Fugl Meyer Assessment, Time Up and Go, 6 Minute Walk Test, 10 Meter Walk Test)
* Clinical measures on lower limb spasticity - Hip, Knee Flexion, Ankle Flexor, Plantar (Modified Ashworth Scale, Modified Tardieu Scale)
* Balance (Berg Balance Scale)
* Pain (Pain Numeric Rating Scale)
* Mood (Hospital Anxiety and Depression Scale)
* FIM
* EQ5D-5L
* Overall length of stay in hospital
* Outcomes events/Complications

Management of adverse events (AEs and SAEs):

At recruitment (Visit 1), patients/ caregivers will be informed to take note and save research coordinator's contact number stated in the ICF. Patients/ caregivers will be reminded to contact research coordinators if patients experience any AE/SAE stated on ICF section 6 from the day of recruitment up to randomization (Visit 2). At randomization (Visit 2) it will again be emphasized to patients and caregivers that they are to continue to monitor for AE/SAE. During the duration of habituation through to the 30-day intervention period, patients/ caregivers are additionally required to report to the study coordinators with regards to any discomfort or issues with the device before proceeding with intervention. During the habituation and the 30-day intervention period, study coordinator will be keeping close contact with the patient/ caregiver by means of messaging apps to ensure compliance to the treatment regime and for AE/SAE reporting.

Patients who are starting the intervention in the inpatient setting will be monitored by the study team for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 21 years old and below 80 years old with a clinically diagnosed first onset ischaemic stroke confirmed by imaging modalities such as computerised tomography (CT) or magnetic resonance imaging (MRI). Previous transient ischemic attack or clinically silent infarct detected by CT/MRI are not considered as previous stroke.
2. Participants within the subacute stage of stroke (Within 14 days from stoke onset)
3. Able to walk with or without assistance
4. Able to understand instructions and give informed consent

Exclusion Criteria:

1. History of craniotomy or placement of implant materials/ device in the body that may affect NIBS including, but not limited to, deep brain stimulator, cardiac implant, cochlear implant
2. Intracranial haemorrhage in the cortical regions
3. History of epilepsy or seizures
4. History of major depression and a history of psychotic disorders
5. Contraindications to tPCS/TENS e.g., pregnancy, presence of skin lesion at the intended treatment areas.
6. Concurrent use of benzodiazepine pyschoactive class of drugs which may affect effects of tPCS
7. Concurrent use of anti-seizure medications (ASMs) which may affect effects of tPCS
8. Presence of significant cognitive impairment/ aphasia rendering patient unable to comply with the treatment protocol
9. Presence of disabling comorbidities that compromises limb function such as orthopaedics or neurological pathologies other than stroke
10. Previous treatments of the lower limb spasticity with botulinum toxin, or alcohol.
11. Prior history of non-invasive brain stimulations

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Portion of Fugl-Meyer Assessment (LE-FMA) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in Lower Extremity Portion of Fugl-Meyer Assessment (LE-FMA).
  Mean change in LE-FMA from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days) and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
Functional Independence Measure (FIM) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in functional independence measured using Functional Independence Measure (FIM) score, in stroke patients with hemiplegia or hemiparesis in the subacute stage.
  Mean change in FIM from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days) and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation +TENS (Control) in lower limb spasticity related to stroke objectively measured using Modified Ashworth scale (MAS).
  Mean change in MAS from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
Modified Tardieu Scale (MTS) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation +TENS (Control) in treatment of lower limb spasticity related to stroke objectively measured using Modified Tardieu Scale (MTS)..
  Mean change in MTS from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
Time Up and Go (TUG) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in walking speed, objectively measured with Time Up and Go (TUG).
  Mean change in TUG from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
10-meter Walk Test (10MWT) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in walking endurance objectively measured with 10-meter Walk Test (10MWT).
  Mean change in 10MWT from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
6-minute Walk Test | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in walking endurance objectively measured using 6-minute Walk Test.
  Mean change in 6-minute Walk Test from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
Berg Balance Scale (BBS) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) in balance objectively measured using Berg Balance Scale (BBS).
  Mean change in BBS from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
Pain Numeric Rating Scale (NRS) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) on pain using pain numeric rating scale (NRS).
  Mean change in NRS from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
EQ5D-5L | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) on quality of life (QOL) measured objectively using EQ5D-5L.
  Mean change in EQ5D-5L from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
Hospital Anxiety Depression Scale (HADS) | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of high frequency tPCS + TENS compared to Sham device stimulation + TENS (Control) on mood using Hospital Anxiety Depression Scale (HADS).
  Mean change in HADS from Visit 1 (Recruitment) to Visit 3 (Last day of intervention, Day 30 post intervention with allowance of + 7 days), and Visit 4 (Final follow-up, Day 90 post intervention with allowance of + 7 days).

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Alexandra Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Time Frame: Beginning 6 months and ending 1 years after the publication of results
Access Criteria: Analyses that qualify for data sharing: meta-analysis Data sharing agreement needs to be signed. Applicant can email the study's Principal Investigator to submit request.

REFERENCES:
- [Background] Kwong PW, Ng GY, Chung RC, Ng SS. Transcutaneous electrical nerve stimulation improves walking capacity and reduces spasticity in stroke survivors: a systematic review and meta-analysis. Clin Rehabil. 2018 Sep;32(9):1203-1219. doi: 10.1177/0269215517745349. Epub 2017 Dec 13. PMID 29232981
- [Background] Kim DY, Lim JY, Kang EK, You DS, Oh MK, Oh BM, Paik NJ. Effect of transcranial direct current stimulation on motor recovery in patients with subacute stroke. Am J Phys Med Rehabil. 2010 Nov;89(11):879-86. doi: 10.1097/PHM.0b013e3181f70aa7. PMID 20962598
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Chib VS, Yun K, Takahashi H, Shimojo S. Noninvasive remote activation of the ventral midbrain by transcranial direct current stimulation of prefrontal cortex. Transl Psychiatry. 2013 Jun 11;3(6):e268. doi: 10.1038/tp.2013.44. PMID 23756377
- [Background] Xueyi Ni, Liru Cui, Ruixia Bi, Jinghua Qian. "Effect of non-invasive brain stimulation on lower limb function in patients after stroke: A PRISMA-compliant systematic review and meta-analysis." Neurology Asia 2021; 26(3) : 501 - 508
- [Background] Julious, S.A. 2010. Sample Sizes for Clinical Trials. Chapman & Hall/CRC. Boca Raton, FL.
- [Background] Dong XL, Sun X, Sun WM, Yuan Q, Yu GH, Shuai L, Yuan YF. A randomized controlled trial to explore the efficacy and safety of transcranial direct current stimulation on patients with post-stroke fatigue. Medicine (Baltimore). 2021 Oct 15;100(41):e27504. doi: 10.1097/MD.0000000000027504. PMID 34731132
- [Background] Zhao W, Wang C, Li Z, Chen L, Li J, Cui W, Ding S, Xi Q, Wang F, Jia F, Xiao S, Guo Y, Zhao Y. Efficacy and safety of transcutaneous electrical acupoint stimulation to treat muscle spasticity following brain injury: a double-blinded, multicenter, randomized controlled trial. PLoS One. 2015 Feb 2;10(2):e0116976. doi: 10.1371/journal.pone.0116976. eCollection 2015. PMID 25643051
- [Background] Wang XB, Chen J, Li TJ, Tao J, Chen LD, He J, Chen LR. [Effect of electroacupuncture in different frequencies on electromyography and ambulation in stroke patients with lower-extremity spasticity: a randomized controlled study]. Zhongguo Zhen Jiu. 2011 Jul;31(7):580-4. Chinese. PMID 21823273
- [Background] Young-Nim Y, Gwang-Cheon P, Myung-Rae C, Min-Yeong S, Chang-Su N, Jae-Young H, Jae-Hong K. Meta-analysis on randomized controlled trials for scalp acupuncture treatment of stroke: A systematic review. J Tradit Chin Med. 2018 Aug;38(4):465-479. PMID 32186072
- [Background] Mogyoros I, Kiernan MC, Burke D. Strength-duration properties of human peripheral nerve. Brain. 1996 Apr;119 ( Pt 2):439-47. doi: 10.1093/brain/119.2.439. PMID 8800939
- [Background] Alon G, Roys SR, Gullapalli RP, Greenspan JD. Non-invasive electrical stimulation of the brain (ESB) modifies the resting-state network connectivity of the primary motor cortex: a proof of concept fMRI study. Brain Res. 2011 Jul 27;1403:37-44. doi: 10.1016/j.brainres.2011.06.013. Epub 2011 Jun 13. PMID 21696709
- [Background] Paneri, B., Khadka, N., Patel, V., Thomas, C., Tyler, W., Parra, L. C., & Bikson, M. (2015). The tolerability of transcranial electrical stimulation used across extended periods in a naturalistic context by healthy individuals (No. e1574). PeerJ PrePrints.
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Plazier M, Joos K, Vanneste S, Ost J, De Ridder D. Bifrontal and bioccipital transcranial direct current stimulation (tDCS) does not induce mood changes in healthy volunteers: a placebo controlled study. Brain Stimul. 2012 Oct;5(4):454-61. doi: 10.1016/j.brs.2011.07.005. Epub 2011 Aug 5. PMID 21962976
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Bernhardt J, Hayward KS, Kwakkel G, Ward NS, Wolf SL, Borschmann K, Krakauer JW, Boyd LA, Carmichael ST, Corbett D, Cramer SC. Agreed definitions and a shared vision for new standards in stroke recovery research: The Stroke Recovery and Rehabilitation Roundtable taskforce. Int J Stroke. 2017 Jul;12(5):444-450. doi: 10.1177/1747493017711816. PMID 28697708
- [Background] Bai X, Guo Z, He L, Ren L, McClure MA, Mu Q. Different Therapeutic Effects of Transcranial Direct Current Stimulation on Upper and Lower Limb Recovery of Stroke Patients with Motor Dysfunction: A Meta-Analysis. Neural Plast. 2019 Nov 16;2019:1372138. doi: 10.1155/2019/1372138. eCollection 2019. PMID 31827495
- [Background] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation for improving spasticity after stroke: A systematic review with meta-analysis. J Rehabil Med. 2016 Jul 18;48(7):565-70. doi: 10.2340/16501977-2097. PMID 27172484
- [Background] Falvey JR, Krafft C, Kornetti D. The Essential Role of Home- and Community-Based Physical Therapists During the COVID-19 Pandemic. Phys Ther. 2020 Jul 19;100(7):1058-1061. doi: 10.1093/ptj/pzaa069. No abstract available. PMID 32302404
- [Background] Satow T, Kawase T, Kitamura A, Kajitani Y, Yamaguchi T, Tanabe N, Otoi R, Komuro T, Kobayashi A, Nagata H, Mima T. Combination of Transcranial Direct Current Stimulation and Neuromuscular Electrical Stimulation Improves Gait Ability in a Patient in Chronic Stage of Stroke. Case Rep Neurol. 2016 Feb 12;8(1):39-46. doi: 10.1159/000444167. eCollection 2016 Jan-Apr. PMID 27293403
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Fang Y, Li J, Liu S, Wang Y, Li J, Yang D, Wang Q. Optimization of electrical stimulation for the treatment of lower limb dysfunction after stroke: A systematic review and Bayesian network meta-analysis of randomized controlled trials. PLoS One. 2023 May 11;18(5):e0285523. doi: 10.1371/journal.pone.0285523. eCollection 2023. PMID 37167257
- [Background] Benowitz LI, Routtenberg A. GAP-43: an intrinsic determinant of neuronal development and plasticity. Trends Neurosci. 1997 Feb;20(2):84-91. doi: 10.1016/s0166-2236(96)10072-2. PMID 9023877
- [Background] Harada A, Teng J, Takei Y, Oguchi K, Hirokawa N. MAP2 is required for dendrite elongation, PKA anchoring in dendrites, and proper PKA signal transduction. J Cell Biol. 2002 Aug 5;158(3):541-9. doi: 10.1083/jcb.200110134. Epub 2002 Aug 5. PMID 12163474
- [Background] Johnson GV, Jope RS. The role of microtubule-associated protein 2 (MAP-2) in neuronal growth, plasticity, and degeneration. J Neurosci Res. 1992 Dec;33(4):505-12. doi: 10.1002/jnr.490330402. PMID 1484385
- [Background] Thibaut A, Russo C, Morales-Quezada L, Hurtado-Puerto A, Deitos A, Freedman S, Carvalho S, Fregni F. Neural signature of tDCS, tPCS and their combination: Comparing the effects on neural plasticity. Neurosci Lett. 2017 Jan 10;637:207-214. doi: 10.1016/j.neulet.2016.10.026. Epub 2016 Oct 17. PMID 27765610
- [Background] Morales-Quezada L, Saavedra LC, Rozisky J, Hadlington L, Fregni F. Intensity-dependent effects of transcranial pulsed current stimulation on interhemispheric connectivity: a high-resolution qEEG, sham-controlled study. Neuroreport. 2014 Sep 10;25(13):1054-8. doi: 10.1097/WNR.0000000000000228. PMID 25055142
- [Background] Morales-Quezada L, Leite J, Carvalho S, Castillo-Saavedra L, Cosmo C, Fregni F. Behavioral effects of transcranial pulsed current stimulation (tPCS): Speed-accuracy tradeoff in attention switching task. Neurosci Res. 2016 Aug;109:48-53. doi: 10.1016/j.neures.2016.01.009. Epub 2016 Feb 3. PMID 26851768
- [Background] Jaberzadeh S, Bastani A, Zoghi M. Anodal transcranial pulsed current stimulation: A novel technique to enhance corticospinal excitability. Clin Neurophysiol. 2014 Feb;125(2):344-51. doi: 10.1016/j.clinph.2013.08.025. Epub 2013 Sep 26. PMID 24074626
- [Background] Dissanayaka T, Zoghi M, Farrell M, Egan G, Jaberzadeh S. The Effects of Monophasic Anodal Transcranial Pulsed Current Stimulation on Corticospinal Excitability and Motor Performance in Healthy Young Adults: A Randomized Double-Blinded Sham-Controlled Study. Brain Connect. 2022 Apr;12(3):260-274. doi: 10.1089/brain.2020.0949. Epub 2022 Feb 16. PMID 34963309
- [Background] Mansouri F, Shanbour A, Mazza F, Fettes P, Zariffa J, Downar J. Effect of Theta Transcranial Alternating Current Stimulation and Phase-Locked Transcranial Pulsed Current Stimulation on Learning and Cognitive Control. Front Neurosci. 2019 Nov 14;13:1181. doi: 10.3389/fnins.2019.01181. eCollection 2019. PMID 31798397
- [Background] Wu Q, Fang G, Zhao J, Liu J. Effect of Transcranial Pulsed Current Stimulation on Fatigue Delay after Medium-Intensity Training. Int J Environ Res Public Health. 2022 Jun 8;19(12):7042. doi: 10.3390/ijerph19127042. PMID 35742289
- [Background] Chamorro-Hinojosa JA, Molina-Rueda F, Carratala-Tejada M. Transcranial Direct Current Stimulation in the Treatment of Gait Disturbance in Post-Stroke Patients: An Overview of Systematic Reviews. Sensors (Basel). 2023 Nov 21;23(23):9301. doi: 10.3390/s23239301. PMID 38067673
- [Background] Li Y, Fan J, Yang J, He C, Li S. Effects of transcranial direct current stimulation on walking ability after stroke: A systematic review and meta-analysis. Restor Neurol Neurosci. 2018;36(1):59-71. doi: 10.3233/RNN-170770. PMID 29439362
- [Background] Guleyupoglu B, Schestatsky P, Edwards D, Fregni F, Bikson M. Classification of methods in transcranial electrical stimulation (tES) and evolving strategy from historical approaches to contemporary innovations. J Neurosci Methods. 2013 Oct 15;219(2):297-311. doi: 10.1016/j.jneumeth.2013.07.016. Epub 2013 Aug 14. PMID 23954780
- [Background] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK; LEAPS Investigative Team. Protocol for the Locomotor Experience Applied Post-stroke (LEAPS) trial: a randomized controlled trial. BMC Neurol. 2007 Nov 8;7:39. doi: 10.1186/1471-2377-7-39. PMID 17996052
- [Background] Robinson CA, Shumway-Cook A, Matsuda PN, Ciol MA. Understanding physical factors associated with participation in community ambulation following stroke. Disabil Rehabil. 2011;33(12):1033-42. doi: 10.3109/09638288.2010.520803. Epub 2010 Oct 5. PMID 20923316
- [Background] Stinear CM, Lang CE, Zeiler S, Byblow WD. Advances and challenges in stroke rehabilitation. Lancet Neurol. 2020 Apr;19(4):348-360. doi: 10.1016/S1474-4422(19)30415-6. Epub 2020 Jan 28. PMID 32004440
- [Background] Kim WS, Cho S, Ku J, Kim Y, Lee K, Hwang HJ, Paik NJ. Clinical Application of Virtual Reality for Upper Limb Motor Rehabilitation in Stroke: Review of Technologies and Clinical Evidence. J Clin Med. 2020 Oct 21;9(10):3369. doi: 10.3390/jcm9103369. PMID 33096678
- [Background] Zhang X, Yue Z, Wang J. Robotics in Lower-Limb Rehabilitation after Stroke. Behav Neurol. 2017;2017:3731802. doi: 10.1155/2017/3731802. Epub 2017 Jun 8. PMID 28659660
- [Background] Sainburg R, Good D, Przybyla A. Bilateral Synergy: A Framework for Post-Stroke Rehabilitation. J Neurol Transl Neurosci. 2013 Oct 23;1(3):1025. PMID 24729985
- [Background] Esht V, Alshehri MM, Balasubramanian K, Sanjeevi RR, Shaphe MA, Alhowimel A, Alenazi AM, Alqahtani BA, Alhwoaimel N. Transcranial direct current stimulation (tDCS) for neurological disability among subacute stroke survivors to improve multiple domains in health-related quality of life: Randomized controlled trial protocol. Neurophysiol Clin. 2024 May;54(3):102976. doi: 10.1016/j.neucli.2024.102976. Epub 2024 Apr 24. PMID 38663043
- [Background] Jagadish A, Natarajan M, Adhia DB, Kuppuswamy A, Guddattu V, Solomon JM. Effect of high-definition transcranial direct current stimulation among late-subacute and chronic stroke survivors with fatigue: A randomized-controlled crossover trial protocol. MethodsX. 2024 Feb 23;12:102629. doi: 10.1016/j.mex.2024.102629. eCollection 2024 Jun. PMID 38435639
- [Background] Duan Q, Liu W, Yang J, Huang B, Shen J. Effect of Cathodal Transcranial Direct Current Stimulation for Lower Limb Subacute Stroke Rehabilitation. Neural Plast. 2023 May 27;2023:1863686. doi: 10.1155/2023/1863686. eCollection 2023. PMID 37274448
- [Background] Youssef H, Mohamed NAE, Hamdy M. Comparison of bihemispheric and unihemispheric M1 transcranial direct current stimulations during physical therapy in subacute stroke patients: A randomized controlled trial. Neurophysiol Clin. 2023 Jun;53(3):102895. doi: 10.1016/j.neucli.2023.102895. Epub 2023 Jul 29. PMID 37517104
- [Background] Tedla JS, Rodrigues E, Ferreira AS, Vicente J, Reddy RS, Gular K, Sangadala DR, Kakaraparthi VN, Asiri F, Midde AK, Dixit S. Transcranial direct current stimulation combined with trunk-targeted, proprioceptive neuromuscular facilitation in subacute stroke: a randomized controlled trial. PeerJ. 2022 Apr 28;10:e13329. doi: 10.7717/peerj.13329. eCollection 2022. PMID 35505681
- [Background] Campanella W, Pedrini R, Vestito L, Marinelli L, Trompetto C, Mori L. Transcranial Direct Current Stimulation in the Treatment of Subacute Post-Stroke Thalamic Aphasia. Eur J Case Rep Intern Med. 2020 Sep 3;7(11):001794. doi: 10.12890/2020_001794. eCollection 2020. PMID 33194851
- [Background] Hsu SP, Lu CF, Lin BF, Tang CW, Kuo IJ, Tsai YA, Guo CY, Lee PL, Shyu KK, Niddam DM, Lee IH. Effects of bihemispheric transcranial direct current stimulation on motor recovery in subacute stroke patients: a double-blind, randomized sham-controlled trial. J Neuroeng Rehabil. 2023 Feb 27;20(1):27. doi: 10.1186/s12984-023-01153-4. PMID 36849990
- [Background] Gong Y, Long XM, Xu Y, Cai XY, Ye M. Effects of repetitive transcranial magnetic stimulation combined with transcranial direct current stimulation on motor function and cortex excitability in subacute stroke patients: A randomized controlled trial. Clin Rehabil. 2021 May;35(5):718-727. doi: 10.1177/0269215520972940. Epub 2020 Nov 23. PMID 33222502
- [Background] NETS Trial Collaboration Group. Efficacy and safety of transcranial direct current stimulation to the ipsilesional motor cortex in subacute stroke (NETS): a multicenter, randomized, double-blind, placebo-controlled trial. Lancet Reg Health Eur. 2024 Jan 2;38:100825. doi: 10.1016/j.lanepe.2023.100825. eCollection 2024 Mar. PMID 38476746
- [Background] Mahmood A, Veluswamy SK, Hombali A, Mullick A, N M, Solomon JM. Effect of Transcutaneous Electrical Nerve Stimulation on Spasticity in Adults With Stroke: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2019 Apr;100(4):751-768. doi: 10.1016/j.apmr.2018.10.016. Epub 2018 Nov 16. PMID 30452892
- [Background] In TS, Jung JH, Jung KS, Cho HY. Effectiveness of Transcutaneous Electrical Nerve Stimulation with Taping for Stroke Rehabilitation. Biomed Res Int. 2021 Aug 25;2021:9912094. doi: 10.1155/2021/9912094. eCollection 2021. PMID 34485529
- [Background] Alon G, Yungher DA, Shulman LM, Rogers MW. Safety and immediate effect of noninvasive transcranial pulsed current stimulation on gait and balance in Parkinson disease. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1089-95. doi: 10.1177/1545968312448233. Epub 2012 May 10. PMID 22581566
- [Background] Liu Z, Dong S, Zhong S, Huang F, Zhang C, Zhou Y, Deng H. The effect of combined transcranial pulsed current stimulation and transcutaneous electrical nerve stimulation on lower limb spasticity in children with spastic cerebral palsy: a randomized and controlled clinical study. BMC Pediatr. 2021 Mar 24;21(1):141. doi: 10.1186/s12887-021-02615-1. PMID 33761932
- [Background] Wang WJ, Zhong YB, Zhao JJ, Ren M, Zhang SC, Xu MS, Xu ST, Zhang YJ, Shan CL. Transcranial pulse current stimulation improves the locomotor function in a rat model of stroke. Neural Regen Res. 2021 Jul;16(7):1229-1234. doi: 10.4103/1673-5374.301018. PMID 33318399
- [Background] Hasenstaub A, Shu Y, Haider B, Kraushaar U, Duque A, McCormick DA. Inhibitory postsynaptic potentials carry synchronized frequency information in active cortical networks. Neuron. 2005 Aug 4;47(3):423-35. doi: 10.1016/j.neuron.2005.06.016. PMID 16055065
- [Background] Jaberzadeh S, Zoghi M. Exploring sensory, motor, and pain responses as potential side or therapeutic effects of sub-2 mA, 400 Hz transcranial pulsed current stimulation. PLoS One. 2023 Dec 13;18(12):e0290137. doi: 10.1371/journal.pone.0290137. eCollection 2023. PMID 38091312
- [Background] Lu Q, Huang G, Chen L, Li W, Liang Z. Structural and functional reorganization following unilateral internal capsule infarction contribute to neurological function recovery. Neuroradiology. 2019 Oct;61(10):1181-1190. doi: 10.1007/s00234-019-02278-x. Epub 2019 Aug 10. PMID 31399852
- [Background] Cassidy JM, Cramer SC. Spontaneous and Therapeutic-Induced Mechanisms of Functional Recovery After Stroke. Transl Stroke Res. 2017 Feb;8(1):33-46. doi: 10.1007/s12975-016-0467-5. Epub 2016 Apr 25. PMID 27109642